CLINICAL TRIAL: NCT06966388
Title: Pilot Study to Evaluate the Feasibility of Twice Daily Use of Topical Azelaic Acid in Breast Cancer Patients Undergoing Radiation
Brief Title: Study to Evaluate the Feasibility of Twice Daily Use of Topical Azelaic Acid in Breast Cancer Patients Undergoing Radiation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-23-20546
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — azelaic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Topical Azelaic Acid (Experimental): Twice daily application of azelaic acid
  Interventions: Drug: Azelaic Acid

INTERVENTIONS:
Drug: Azelaic Acid — A thin layer of Azelaic acid should be applied to the entire area of radiation treatment twice daily, each day of the week (including weekends) starting one week prior to the start of radiation, then during the entire course of radiation treatment (usually 3-5 weeks), and for 3 weeks following the completion of radiation treatment.

SUMMARY:
This pilot study will evaluate the feasibility of at least twice daily use of azelaic acid in breast cancer patients undergoing radiation treatment.

DETAILED DESCRIPTION:
Patients will use azelaic acid twice daily (morning and evening) beginning 1 week before radiation treatment, and will continue use until 3 weeks after completion of radiation treatment

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

* Self-reports as Black, Asian, Hispanic/Latin, ethnically originating from the Mediterranean rim or Pacific rim, or she/he tans easily in the sun
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2 (Appendix 1, Section 18)
* Attestation by the patient that she/he is not pregnant, lactating, or planning to become pregnant, or planning to father a baby during the study period
* Histologic confirmation of breast malignancy (with TNM staging) If the patient did not receive adjuvant chemotherapy, adjuvant radiation must start within 180 days of lumpectomy or mastectomy. If the patient received adjuvant chemotherapy, adjuvant radiation should start within 60 days of the last dose of chemotherapy
* Treatment plan includes one of the following:

  * Conventionally fractionated whole breast radiation (45-50 Gray in 25 fractions)
  * Moderately hypofractionated whole breast radiation (42.56 Gray in 16 fractions or 40 Gray in 15 fractions)
  * Conventionally fractionated chest wall radiation (45-50 Gray in 25 fractions)
  * Partial breast radiation (42.56 Gray in 16 fractions, 40 Gray in 15 fractions, or 30 Gray in 5 fractions) if using 3D conformal radiation or if the tumor is located close to the skin surface
* Treatment of the regional lymph nodes, a tumor bed boost (4-8 fractions), and use of tissue-equivalent bolus on the chest wall may be included at the discretion of the treating physician.
* Radiation will be photon-based. Note: If the patient receives a boost, photons and/or electrons may be used at the discretion of the treating physician.

Exclusion Criteria:

* Prior radiotherapy to any portion of the planned treatment site
* Current inflammatory breast cancer or gross dermal involvement at initiation of radiotherapy
* Concomitant immunotherapy or cytotoxic chemotherapy. Concomitant HER2 directed therapy or concomitant endocrine therapy is allowed
* Active rash or dermatitis within the treatment field, or a history of any rash or dermatologic condition within the treatment field
* Active collagen vascular diseases (ie lupus erythematosus, scleroderma, dermatomyositis)
* History of organ transplant or bone marrow transplant
* History of hypersensitivity or allergic reaction to any ingredients in the topical azelaic acid formulation
* Has used within 28 days prior to baseline:

  * topical retinoids to the breast
  * oral retinoids
  * systemic (oral or injectable) antibiotics known to have an impact on the severity of skin rash or sun-sensitivity (eg, containing tetracycline and its derivatives, erythromycin and its derivatives, sulfamethoxazole, or trimethoprim)
  * systemic corticosteroids or immunosuppressive drugs, except as part of standard chemotherapy treatment or used for an IV contrast allergy
* Has used on treated breast within 2 weeks prior to baseline:

  * topical corticosteroids
  * topical antibiotics
  * topical medications for skin rash (eg, metronidazole, azelaic acid)
* Radiation therapy will be proton therapy or carbon therapy
* External beam partial breast irradiation, brachytherapy partial breast irradiation, or intraoperative radiation are included in the treatment plan Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Determine the feasibility of twice daily use of topical azelaic acid in patients undergoing breast radiation therapy | One week prior to radiation treatment, daily during radiation treatment up to 5 weeks, three weeks following radiation treatment
  The percentage of days patients used azelaic acid at least once.

SECONDARY OUTCOMES:
Evaluate patient-reported tolerability of topical azelaic acid | Weekly during radiation treatment, and Up to three weeks following radiation treatment
  The percentage of patients that self report adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Todd C. Adams, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No